CLINICAL TRIAL: NCT02933086
Title: An Intervention Program for the Trunk Neuromuscular Pattern and Postural Control in Pregnant With Low Back Pain: A Feasibility and Clinical Trial Study
Brief Title: An Intervention Program for the Trunk Neuromuscular Pattern and Postural Control in Pregnant With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Rubens Alexandre da Silva Jr, Titular professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.579.189
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pregnancy Complications; Low Back Pain
Keywords: Pregnant; Low Back Pain; Postural Control
MeSH Terms: conditions — Pregnancy Complications; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G1: exercises for lumbar stabilization (Experimental): G1, will perform therapy with specific exercises for lumbar stabilization including the Swiss ball as therapeutic resource
  Interventions: Other: Specific exercises for lumbar stabilization
- G2: conventional therapy (Experimental): G2, will perform conventional therapy including stretching of lower limbs and trunk.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Specific exercises for lumbar stabilization — The Group 1 (G1) will perform therapy with specific exercises for lumbar stabilization whith the Swiss ball as a therapeutic resource, including warming; stretching of hamstrings, paraspinals, trapezes; phasic perineal exercise; tonic perineal exercise; pelvic lumbar synergism; trunk mobility; mobility of the shoulder girdle; balance; and slow pelvic balance.
  Arms: G1: exercises for lumbar stabilization
Other: Conventional therapy — The Group 2 (G2) will perform conventional therapy including stretching of lower limbs and trunk, with passive stretching of hamstrings; gluteus maximus; piriform; paraspinals; lumbar square; latissimus dorsi; scalene; trapezius.
  Arms: G2: conventional therapy

SUMMARY:
The relevance of this study is given by the feasibility to assess the effect of an intervention program based on the functionality and trunk neuromuscular activity and postural control in pregnant women with low back pain. The main outcomes will be computed by electromyography measurement so that to assess the trunk neuromuscular activation pattern as well as by force platform parameters for determining of postural control. Clinical symptoms such as pain intensity, perception of disability and fear and avoidance will also be computed. This is the first study to compare two intervention methods using the main biological outcomes related to trunk segment function.

DETAILED DESCRIPTION:
For this study, a proposal of a 6-week intervention program will be carried out with lumbar stabilization exercises and clinical orientations, on 20 low back pregnant patients recruited by convenience and voluntaries from the community. Before intervention, all participantes will be evaluated by: electromoyography during three exercises, balance, and clinical outcomes such as pain, disability and psychological factors. All baseline testing and evaluation will be performed by a blinded evaluator to the study intervention.

Afterwards, the participants will be randomized in two groups by a blinded evaluator (people not enroled to study): G1: exercises for lumbar stabilization; and G2: conventional therapy.

The intervention will follow six weeks, with 50 minutes of duration each session of therapy including measurement of blood pressure, heart rate and the Visual Analogue Scale (VAS) before and after each session, and the perception of exercise intensity monitored by Borg Scale. Within this proposal, the exercise sessions will be twice a week, lasting 40 minutes each, and followed by 10 minutes of theoretical orientation. The intervention will follow the CONSORT recommendations for randomized controlled trials. The intervention will start in: G1 (n=10), which will perform therapy with specific exercises for lumbar stabilization including the Swiss ball as therapeutic resource; while G2 (n=10, control group) will perform conventional therapy including stretching of lower limbs and trunk. The participants will not be blind to the study due to the characteristic of the exercises that often reflect to the improvement of the symptoms. In case of eventual losses, the intention-to-treat method will be used for the analyses.

After the intervention, all groups will be invited to come back to the laboratory to proceed the same evaluation from baseline (trunk activation during three exercises, balance, and clinical outcomes) For the analysis two-way ANOVA with repeated measures will be performed to compare the effects of the intervention (two groups) and times (baseline vs. end 6-weeks measurement)the effects of interaction (Groups x Times).

ELIGIBILITY:
The inclusion criteria were:

* Have between 19-29 weeks of pregnancy;
* Have performed prenatal clinical monitoring;
* Have chronic low back pain (> 3 months) without irradiation for knees.
* Not being under medication or physical therapy treatment for low back pain in the last three months;
* To be able to perform physical activity consistent to the pregnancy;
* To present normal conditions of responsiveness, cognition and speaking;
* To be voluntary.

The exclusion criteria were:

* Signs or symptoms of other pathology including coexisting pathology, a recent history (within 3 months) of surgery in the locomotor system;
* Respiratory, neurological or cardiovascular diseases.
* Several musculoskeletal disorders.
* Limitations for physical exercise.
* Allergic reaction to adhesive tape,

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Eletromyography measurement | Change from baseline muscular activation at 6 weeks
  Level of muscular activaity of trunk from eletromyography surface processing.

SECONDARY OUTCOMES:
Force platform measurement | Change from baseline balance performance at 6 weeks
  Force platform measurement during balance performance using centre of pressure measures to assess balance performance.

OTHER OUTCOMES:
Visual Analogic Scale | Change from baseline pain intensity at 6 weeks.
  Pain measurement using Short Version of Pain Questionnaire Mc Gill and Visual Analogue Scale (VAS).
Disability questionnaire | Change from baseline disability status at 6 weeks.
  Disability measurement using Roland Morris questionnaire.
Fear-avoidance questionnaire | Change from baseline Fear-avoidance status at 6 weeks.
  Fear-avoidance model measurement using Waddel questionnaire related to work and physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens A da Silva Jr., Phd, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Laboratory of Functional Assessment and Human Motor Performance (LAFUP), Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Keeffe M, O'Sullivan P, Dankaerts W, O'Sullivan K. Swiss ball enhances lumbar multifidus activity in chronic low back pain: A letter to the editor. Phys Ther Sport. 2015 May;16(2):202-3. doi: 10.1016/j.ptsp.2015.03.001. Epub 2015 Mar 11. No abstract available. PMID 25840522
- [Background] Liddle SD, Pennick V. Interventions for preventing and treating low-back and pelvic pain during pregnancy. Cochrane Database Syst Rev. 2015 Sep 30;2015(9):CD001139. doi: 10.1002/14651858.CD001139.pub4. PMID 26422811
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Madeira HG, Garcia JB, Lima MV, Serra HO. [Disability and factors associated with gestational low back pain]. Rev Bras Ginecol Obstet. 2013 Dec;35(12):541-8. doi: 10.1590/s0100-72032013001200003. Portuguese. PMID 24500508